CLINICAL TRIAL: NCT05971043
Title: Skin Disorders in Patients Using Methamphetamine
Brief Title: Skin Disease in Methamphetamine Abuse
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa mohamed hafez, principal investigator Dr asmaa mohamed hafez, Assiut University
Other Study IDs: meth addiction
Record Dates: First submitted 2023-07-09; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Methamphetamine Abuse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. To detect the skin diseases in patients using methamphetamine

DETAILED DESCRIPTION:
Methamphetamine is a stimulant drug that associated with a broad spectrum of health conditions, include addiction, mental health disorders, and overdose. The Drug Enforcement Agency (DEA) classifies it as a Schedule II drug. This means that the drug has a high potential for misuse. The drug is also called crystal meth, ice, and blue.

Methamphetamine use has increased in Egypt especially in upper Egypt. Literature on cutaneous manifestations among methamphetamine users is limited, although cellulitis, delusion of parasitosis (DOP), hyperhidrosis, formication and prurigo nodularis (PN) have been attributed to methamphetamine users. While the relationship between skin lesions and substance use in not fully defined, there is some evidence that points to the development of these itchy, red lesion also known as meth sore after meth use. Meth sores often look like small round red patches on your skin, they can often be confused with acne when they appear on the face or a rash when they appear on other parts of the body.

Meth sores form as a result of heavy meth misuse. other signs of meth abuse at the stage where sores likely to develop include:

* Weight loss
* Paranoia
* Hallucinations
* Aggressive behavior
* Being easily distracted
* Tooth and gum decay
* Changes in brain structure

ELIGIBILITY:
Inclusion Criteria:

* Patients using methamphetamine

Exclusion Criteria:

* 1. Pregnant and lactating patients. 2. Patients with chronic diseases

Ages: 14 Years to 75 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: cross-sectional, questionnaire-based, study including clinical assessment of diseases severity.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-08-03 (Estimated); Primary Completion 2024-08-20 (Estimated); Study Completion 2024-09-20 (Estimated)

PRIMARY OUTCOMES:
skin disorders in patients using methamphetamine | baseline
  questionnaire-based study To detect the skin diseases and manifestation appears in patients using methamphetamine

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Shawkey gomaa, Lecturer, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barnes AJ, Smith ML, Kacinko SL, Schwilke EW, Cone EJ, Moolchan ET, Huestis MA. Excretion of methamphetamine and amphetamine in human sweat following controlled oral methamphetamine administration. Clin Chem. 2008 Jan;54(1):172-80. doi: 10.1373/clinchem.2007.092304. Epub 2007 Nov 2. PMID 17981924